CLINICAL TRIAL: NCT04848428
Title: Feasibility and Preliminary Effects of a Tailored Web-based Mindfulness-based Intervention to Prevent Chronic Pain After Major Surgery
Brief Title: Online Mindfulness-based Intervention to Prevent Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Geraldine Martorella, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 046073
Record Dates: First submitted 2021-04-07; First posted 2021-04-19 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Pain, Postoperative; Chronic Pain; Pain Catastrophizing; Pain, Acute
Keywords: postoperative pain; mindfulness; chronic pain
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain; Acute Pain

STUDY DESIGN:
Intervention Model Description: 2-arm pilot RCT
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Mindfulness-based intervention (Experimental): Four weekly sessions are planned. The first session will focus on providing feedback regarding post-surgical pain. The second session will focus on teaching mindfulness strategies. The third session will focus on practicing one of the two strategies. Of note, sessions 2 and 3 will start with cognitive restructuring strategies. The 4th session consists in a booster providing feedback and reminders about cognitive reactions to pain and mindfulness meditation. The participants will be asked to practice meditation 5 days a week, for a total of 4 weeks
  Interventions: Behavioral: Online mindfulness-based cognitive therapy
- Online standardized education (Active Comparator): In addition to usual care, the CG will have access to one 15-minute standardized educational online session on persistent post-surgical pain, how pain and stress may interact and their potential impact on recovery.
  Interventions: Behavioral: Online standardized education

INTERVENTIONS:
Behavioral: Online mindfulness-based cognitive therapy — The first session will first focus on providing feedback regarding post-surgical pain. The second session will focus on teaching mindfulness strategies. The third session will focus on practicing one of the two strategies. Of note, sessions 2 and 3 will start with cognitive restructuring strategies for the moderate-high risk profile patients. The 4th session consists in a booster providing feedback and reminders about cognitive reactions to pain and mindfulness meditation. The participants will be asked to practice meditation 5 days a week, for a total of 4 weeks
  Other Names: Online MBCT
  Arms: Online Mindfulness-based intervention
Behavioral: Online standardized education — One 15-minute educational session on postoperative pain, the relationship between pain, thoughts and emotions and brief overview of strategies.
  Arms: Online standardized education

SUMMARY:
Cardiac and orthopedic surgeries are frequent procedures. However, pain after a major surgery may become chronic (lasting >3 months) in adults. Once discharged from the hospital, patients are at risk for chronic post-surgical pain (CPSP) and prolonged opioid use, as they become isolated with high levels of pain. Psychological risk and protective factors such as pain-related catastrophic thoughts and pain acceptance will determine their ability to cope and their opioid use, which makes a support for pain self-management crucial. There is limited research on psychological interventions for pain in the subacute/rehabilitation phase after major surgery. Further, these interventions are demanding and not tailored. Previous work from the Principal Investigator in the acute/hospitalization phase shows that a brief, Web-based intervention tailored to modifiable psychological factors may modulate these and reduce postoperative pain interference. Recently, studies on mindfulness-based cognitive therapy (MBCT) have multiplied regarding their potential effect on pain acceptance and catastrophic thoughts. Brief, Web-based MBCT for the prevention of CPSP have not been examined. Therefore, a pilot test of a 4-week tailored, Web-based MBCT intervention for adults in the rehabilitation phase will be conducted by 1) assessing the acceptability/feasibility of the intervention; and 2) examining preliminary effects on pain intensity and pain interference with activities, as well as pain acceptance and catastrophic thoughts. This research is significant because it targets the trajectory of CPSP, a leading cause of disability and opioid misuse. This approach is innovative because it promotes pain self-management through the modulation of individual factors. If successful, the intervention could be expanded to numerous populations at risk for chronic pain.

DETAILED DESCRIPTION:
A single blinded pilot randomized controlled trial will be used to assess preliminary efficacy of the Web-based MBCT intervention following major surgery (Coronary Artery Bypass Grafting [CABG] or/and Valve Replacement [VR]; Total knee or hip replacement). An experienced research assistant (RA) will be responsible of participants' recruitment and informed consent procedures at the time of follow-up (usually 2 weeks after surgery). The study will be advertised on the rehabilitation units and surgeon's offices with posters and flyers . If interested, clinical team will contact the RA and inclusion criteria will be assessed. After having collected baseline measures, participants will be randomized into two groups by the principal investigator (PI): one receiving both the 4-week Web-based MBCT intervention and the usual care procedure (Experimental Group: EG), the other one receiving solely one standardized educational online session and the usual care procedure (Control Group: CG). Participants from the CG will be given the opportunity to receive the entire intervention once the study will be completed.

Permuted-block randomization with an allocation ratio of 1:1 will be used to generate a list through computer software. The list and envelopes will be prepared by a PI's colleague who will not be involved in this study. The RA who will be responsible of the entire data collection will be blinded to patient group assignment.

All participants will complete baseline measures via a telephone interview or a Qualtrics® survey (T0). Usual socio-demographic variables --i.e., age, sex, civil status, living conditions, education level, and employment status will be assessed. Considering the reciprocity between pain and, anxiety and depression, measures will be taken with the PHQ-4 before intervention (T0), and after intervention (T1). Presence of chronic pain before surgery will be documented as well. Analgesic medication intake will be documented at all time points. The protocol will favor an intention-to-treat approach for the analysis of results. Participants' flow will be reported according to the CONSORT guidelines for psychological interventions. Student's t-tests or chi-square tests will be performed for each socio-demographic, medico-surgical and baseline psychological variables to assure that equivalence of groups was obtained through randomization, although this procedure is not mandatory. The statistical analysis will be mostly descriptive (mean, standard deviation for continuous outcomes and, frequency and proportion for categorical outcomes) with 95% confidence intervals when appropriate. Pain intensity, pain interference, mindfulness, pain acceptance, pain-related catastrophic thoughts, and psychological well-being scores will be summarized using descriptive statistics presented per group at each time point. Further, treatment effect will be estimated and presented with 95% CI at each time point. A first set of exploratory analysis will be carried out to compare the evolution of pain intensity, pain interference, mindfulness, pain acceptance, pain-related catastrophic thoughts, and psychological well-being in each group through the use of two-way ANOVA with repeated measures (pre-intervention, post-intervention). A second set of analyses will assess the impact of the intervention on the prevalence and severity of CPSP (pain intensity and interference, mindfulness, pain acceptance, pain-related catastrophic thoughts, and psychological well-being). Repeated measures ANOVA and repeated measures logistic regression will be performed to compare groups for illustrative purposes since the study is not powered to show statistical significance. An alpha level of significance of 0,05 will be used for all analyses. If interactions are found (p<0,05), post-hoc comparisons will be performed. Lastly, qualitative data obtained from individual interviews will be content analyzed.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* first-time elective CABG and/or VR via a median sternotomy OR total knee or hip replacement
* presence of pain at movement ≥4/10
* ability to understand and complete questionnaires in English
* ability to use an electronic device such as a smartphone, computer or tablet

Exclusion Criteria:

- unable to consent because of physical or mental incapacity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline Pain Intensity after intervention | pre-intervention, immediately after the intervention
  0-10 Numerical Rating Scale (Brief Pain Inventory)
Change from baseline Pain interference after intervention | pre-intervention, immediately after the intervention
  0-10 Numerical Rating Scale (Brief Pain Inventory) several daily activities such as housework, sleep, etc

SECONDARY OUTCOMES:
Change from Baseline Mindfulness after intervention | pre-intervention, immediately after the intervention
  The Cognitive and Affective Mindfulness Scale-Revised (CAMS-R): 12-item scale This scale captures the broad concept of mindfulness according to 4 domains (attention, present focus, awareness, acceptance/non-judgement) without being specific to any particular meditation or strategy.
Change from baseline Chronic pain acceptance after intervention | pre-intervention, immediately after the intervention
  Chronic Pain Acceptance Questionnaire (CPAQ-8): 8-item scaleThis scale comprises two subscales: the degree to which patients engage in daily living activities regardless of pain (4 items), and the willingness to experience pain (4 items).
Change from Baseline Pain catastrophizing after intervention | pre-intervention, immediately after the intervention
  The Pain Catastrophizing Scale (PCS) includes 13 items and will be used to assess patients' pain-related catastrophic thoughts. It includes 13 items divided into three subscales: rumination (4 items), magnification (3 items) and helplessness (6 items). Each item is rated on a 5-point scale with the end points "not at all" (0) and "all the time" (4).

OTHER OUTCOMES:
Patient perception of the intervention's effectiveness, appropriateness, suitability and willingness to adhere | immediately after intervention
  The intervention acceptability will be rated using the Treatment Acceptability and Preferences (TAP) questionnaire which consists in a 5-point Likert scale regarding four attributes: 1) appropriateness in helping patients manage pain, 2) effectiveness in promoting pain management, 3) suitability and, 4) willingness to adhere, with the use of the Treatment Acceptability and Preference (TAP) measure.The ratings refer to a 5-point scale ranging from not at all (0) to very much (4). Additionally,thirty-minute semi-structured individual interviews (telephone or videoconference) will be then conducted by the RA. Patients' rating of each component will be used to solicit feedback on the intervention's acceptability and on the need for further modifications. Interviews will be digitally recorded and transcribed by a trained RA.
Incidence of refusal and dropout | during the intervention, through study completion (1 month)
  percentages of refusal and dropout as well as reasons will be reported
Treatment dosage | during the intervention, immediately after intervention, through study completion (1 month)
  percentages of participants completing the sessions according to the planned schedule will be assessed through Website monitoring
Treatment adherence | during the intervention, immediately after intervention, through study completion (1 month)
  number of times the sessions were accessed by participants

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine Martorella, PhD, Principal Investigator — Florida State University
Locations (1):
- Tallahassee Memorial Hospital, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided